CLINICAL TRIAL: NCT05636514
Title: A Phase I Study of Oral Decitabine and Cedazuridine (ASTX727) In Combination With Defactinib (VS-6063) as Therapy of Myelodysplastic Syndromes and Low-blast Acute Myeloid Leukaemia
Brief Title: Combined Evaluation of Epigenetic and Sensitising Therapy in AML and MDS
Acronym: CELESTIAL-MDS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Clinical Hub for Interventional Research (CHOIR) (Other Government)
Collaborators: The University of New South Wales (Other); Australian National University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-M-002
Record Dates: First submitted 2022-11-01; First posted 2022-12-05 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Myelodysplastic Syndromes; Chronic Myelomonocytic Leukemia; Acute Myeloid Leukemia
Keywords: Myelodysplastic Syndromes; Chronic Myelomonocytic Leukemia; Acute Myeloid Leukemia; MDS; AML; CMML
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Acute | interventions — Decitabine; cedazuridine; decitabine and cedazuridine drug combination; defactinib

STUDY DESIGN:
Intervention Model Description: A phase 1, open-label, 3+3 dose escalation, multicentre study. All participants will receive a fixed dose of ASTX727, with escalation and de-escalation of the dose of defactinib. Enrolled participants will receive one cycle of ASTX727 alone (pre-phase) followed by five cycles of ASTX727 in combination with defactinib (combination phase). Participants with stable or responding disease by IWG criteria will be eligible to proceed to a continuation phase of monotherapy with ASTX727.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Decitabine/cedazuridine + defactinib (Experimental): Decitabine/cedazuridine taken days 1-5 of each 28 day treatment cycle, cycle 1 to 6
  Defactinib taken on days 1-5 of each 28 treatment day cycle from cycle 2 to cycle 6.
  Interventions: Drug: Decitabine/Cedazuridine 35 Mg-100 Mg ORAL TABLET; Drug: Defactinib

INTERVENTIONS:
Drug: Decitabine/Cedazuridine 35 Mg-100 Mg ORAL TABLET — Fixed dose treatment cycles 1 to 6. Cycle 1 is monotherapy, cycles 2 to 6 combination therapy with defactinib.
  Other Names: ASTX727; INQOVI
Drug: Defactinib — Defactinib treatment will commence with at the starting dose (dose level 1) from cycle 2 to 6.
  Dose escalation/de-escalation will proceed based on the MTD determination.
  Dose Level 1: 200mg Defactinib twice daily (starting dose level)
  Dose Level 2: 400mg defactinib twice daily
  Dose Level -1: 200mg Defactinib daily
  Other Names: VS-6063

SUMMARY:
The goal of this project is to see if two new potential treatments (defactinib and the combination tablet of decitabine/cedazuridine) can safely be combined to improve outcomes in people with high-risk myelodysplastic syndrome (MDS), certain forms of Acute Myeloid Leukaemia (AML), and Chronic Myelomonocytic Leukaemia (CMML). Decitabine/cedazuridine is approved for use by the Australian Therapeutics Goods Administration (TGA) as treatment for MDS. Defactinib is an experimental treatment. This means it is not an approved treatment for MDS in Australia. So far it has been given to over 625 patients in studies across the world.

All study participants will receive active treatment, there is no placebo. Participants will take the decitabine/cedazuridine treatment once a day for 5 days in a row (day 1 to day 5) on its own for the first month (cycle). From month 2 participants will take the decitabine/cedazuridine treatment and will also take the defactinib treatment, both for 5 days in a row on days 1 to day 5 each month (cycle). Defactinib is taken twice a day.

DETAILED DESCRIPTION:
The primary objective of this study is to establish the maximum tolerated dose of the combination of ASTX727 (decitabine/cedazuridine) and defactinib administered for 5 days of a 28-day cycle in participants with high-risk MDS, low-blast Acute Myeloid Leukaemia (AML), or Chronic Myelomonocytic Leukaemia (CMML). The secondary objectives are to gather in vivo evidence that adjuvant focal adhesion kinase (FAK) inhibition promotes HSPC mobilisation and proliferation, increased decitabine (DAC) incorporation and DNA hypomethylation in bone marrow and peripheral blood mononuclear cells (MNCs) and increased hematopoietic output from haematopoietic stem and progenitor cells (HSPCs) {colony forming unit-cells [CFU-Cs]}) when used in combination with ASTX727. DAC incorporation and global DNA hypomethylation in peripheral blood and bone marrow MNCs will be assayed longitudinally using a mass spectrometry method (AZA-MS) and cell cycle changes in bone marrow MNCs using a flow cytometry method, which were both developed by these investigators.

Data from previous studies conducted by these Investigators, has shown that hypomethylating agents (HMA) do not alter the clonal architecture of mutant HSPCs but increase their hematopoietic output by epigenetic means. To demonstrate that adjuvant decitabine promotes HMA induced changes in mutant HSPCs, the investigators will use a method adapted from Rand and Molloy, and improved by this research group, for use in single cells in combination with simultaneous assessment of mutations and gene expression. Given the known impact of FAK inhibition on stromal and immune cells in the tumor microenvironment, the investigators will also assess longitudinal changes in these components using single cell transcriptomics and mass cytometry. Along with clinical efficacy data, the investigators will assess pre- and post-treatment density of mutant clones by sequencing a panel of genes associated with myeloid malignancies.

This study's overarching aim is to assess whether defactinib can be safely combined with ASTX727 to improve clinical outcomes in patients with high-risk MDS, low blast AML and CMML. This study will also provide correlative data to support the underlying hypothesis for use of this combination to optimise future HMA therapy.

Treatment of participants will occur in three phases: an initial 'prephase' cycle of monotherapy with ASTX727 (decitabine/cedazuridine) day 1 to 5 of a 28 day cycle (Cycle 1); a combination phase of up to 5 28 day cycles of ASTX727 (decitabine/cedazuridine) in combination with defactinib (VS-6063) (Cycles 2 through 6); and a continuation phase of monotherapy with ASTX727 decitabine/cedazuridine in participants continuing to derive benefit. Participants may continue therapy in continuation phase until progressive disease or the development of unacceptable toxicity.

Adverse events during the first combination cycle (Cycle 2) will be assessed to determine the maximum tolerated dose (MTD) for combination ASTX727 (decitabine/cedazuridine) with defactinib (VS-6063).

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria at the time of screening:

1. Age ≥ 18 years
2. Documented diagnosis of:

   1. Myelodysplastic syndrome (MDS) classified as intermediate-2 or high risk according to the International Prognostic Scoring System (IPSS), or
   2. Acute Myeloid Leukaemia (AML) with 20-30% marrow blasts and multilineage dysplasia, according to WHO classification, or
   3. Chronic myelomonocytic leukemia (CMML) with 10-29% marrow blasts without myeloproliferative disorder according to World Health Organisation (WHO) classification. This confirmation will be from either the Bone marrow aspirate (BMA) performed at screening or a standard of care BMA if performed up to 6 weeks before cycle 1 day 1.
3. Performance status by Eastern Cooperative Oncology Group (ECOG) Criteria of 0 or 1
4. Unsuitable for allogeneic stem cell transplantation
5. For participants who were born female who are of childbearing potential (FCBP) the following criteria apply:

   1. Agreement to use at least two highly effective (per Clinical Trial Facilitation Group) contraceptive methods throughout the study, and for 6 months following the last dose of study drug:

      * Oral/intravaginal/transdermal combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation
      * Oral/injectable/implantable progestogen-only hormonal contraception associated with inhibition of ovulation
      * Intrauterine device (IUD)
      * Intrauterine hormone-releasing system (IUS)
      * Bilateral tubal occlusion
      * Vasectomised partner
      * Sexual abstinence and
   2. Confirmation of a negative serum pregnancy test at screening.
6. Male participants with a partner who was born female and is of childbearing potential must agree to use at least two highly effective (per Clinical Trial Facilitation Group) contraceptive methods throughout the course of the study and for 6 months following the last dose of study drug, and refrain from donating sperm during the same period
7. Provision of signed written informed consent document prior to any study related assessments or procedures being carried out.

Exclusion Criteria:

Participants who meet any of the following criteria at the time of screening/enrolment (up to 28 days prior to Cycle 1 Day 1) will be ineligible for entry into the study:

1. Acute myeloid leukemia (AML) with ≥ 30% blasts in bone marrow according to WHO classification.
2. Prior allogeneic or autologous stem cell transplant.
3. Prior receipt of >1 cycle of a hypomethylating agent.
4. Clinical evidence of central nervous system (CNS) or pulmonary leukostasis, disseminated intravascular coagulation, or CNS leukemia.
5. Use of any of the following within 28 days prior to cycle 1 day 1:

   1. thrombopoiesis-stimulating agents ([TSAs]; eg, Romiplostim, Eltrombopag, Interleukin-11)
   2. ESAs (Erythropoiesis stimulating agent) and other RBC (Red blood cell) hematopoietic growth factors (eg, interleukin-3)
   3. Any other investigational medicinal product from another clinical trial.
6. Exposure to any medication, supplement, traditional/herbal medicine, or food with potential for drug-drug interactions with defactinib during the course of the study. This includes:

   1. strong CYP3A4 inhibitors or inducers
   2. strong CYP2C9 inhibitors or inducers
   3. P-glycoprotein (P-gp) inhibitors or inducers
7. Treatment with warfarin. Patients on warfarin can be converted to low molecular-weight heparin or direct oral anticoagulants (DOACs). Participants unwilling or unable to convert to an alternative are not eligible.
8. Use of hydrea for more than 7 days prior to cycle 1 day 1. Use within that time period is permissible.
9. Concurrent use of corticosteroids unless the participant is on a dose of ≤10mg prednisolone or equivalent for medical conditions other than MDS.
10. Active inflammatory bowel disease, or any other gastrointestinal disorder or defect that would interfere with the ingestion, absorption, distribution, metabolism or excretion of the investigational products and/or predispose the participant to an increased risk of gastrointestinal toxicity.
11. Prior history of malignancies, other than MDS unless the participant has been free of the disease for ≥ 12 months. However, participants with the following history/concurrent conditions are allowed:

    1. Basal or squamous cell carcinoma of the skin
    2. Carcinoma in situ of the cervix
    3. Carcinoma in situ of the breast
    4. Incidental histologic finding of prostate cancer (T1a or T1b using the tumor, nodes, metastasis [TNM] clinical staging system)
12. Significant active cardiac disease within the previous 6 months, including:

    1. New York Heart Association (NYHA) class III or IV congestive heart failure;
    2. Unstable angina or angina requiring surgical or medical intervention; and/or
    3. Myocardial infarction
13. Baseline Qt interval greater than 440 milliseconds (males) or 450 milliseconds (females)
14. Active systemic infection:

    1. Infection with ongoing signs/symptoms related to the infection without improvement despite appropriate anti- infectives
    2. Active Hepatitis B (HBV) infection (defined as HBsAg positive, or HBcAb positive and measurable HBV DNA; participants who are HBcAb positive must have HBV DNA assayed during screening)
    3. Participants with Human Immunodeficiency Virus (HIV) or Hepatitis C (HCV) infection will be considered individually by the coordinating principal investigator:

       * Those with HIV will generally be eligible if receiving antiretroviral therapy, HIV viral load (VL) is suppressed <50 copies/mL , and CD4≥350 cells/mm3.
       * Those with HCV will generally be eligible if there is no evidence of clinical hepatic dysfunction or other systemic manifestations of HCV disease and the hepatic parameters below are met. Consideration should be given to curative HCV therapy prior to enrollment in consultation with HCV clinician, if possible.
15. Any of the following laboratory abnormalities:

    1. Serum AST/SGOT (Aspartate transaminase / Serum glutamic oxaloacetic transaminase) or ALT/SGPT (Alanine aminotransaminase / Serum glutamic pyruvate transaminase) > 2.5 x ULN (upper limit of normal)
    2. Serum total bilirubin > 1.5 x ULN. Patients with Gilbert syndrome may enroll if total bilirubin < 51 umol/L upon discussion with the coordinating investigator
    3. Evidence of autoimmune hemolytic anemia manifested as a corrected reticulocyte count of > 2% with either a positive direct anti-globulin test (DAT) or over 50% of indirect bilirubin
    4. Creatinine clearance <50 ml/minute as calculated by the CockcroftGault formula or serum creatinine of ≥ 1.5 x ULN.
    5. Absolute WBC (white blood cell count) ≥ 20 x 109/L f ) Participants with isolated individual lab abnormalities considered to be disease related will be considered individually in consultation with the Coordinating Principal Investigator.
16. Known or suspected hypersensitivity to study drugs or their constituents.
17. Pregnant or breast-feeding.
18. Any condition not already outlined above which, in the opinion of the clinical investigator, would place the participant at risk if they participated or would jeopardise adherence or follow up or confound the ability to interpret study data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-12-14 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | Once 3 participants have completed 2 cycles, assessed at approximately 2 months (each cycle is 28 days)
  Maximum dose at which no more than 1 of 6 participants experience a dose limiting toxicity (DLT)

SECONDARY OUTCOMES:
Number of Grade 3 or 4 adverse events | End of cycle 6 (24 weeks, each cycle is 28 days)
  Number of participants experiencing Grade 3 or 4 adverse events or serious adverse events (SAEs) during cycles 1-6, along with description of events
Proportion of Grade 3 or 4 adverse events | End of cycle 6 (24 weeks, each cycle is 28 days)
  Proportion of participants experiencing Grade 3 or 4 adverse events or serious adverse events (SAEs) during cycles 1-6, along with description of events
Number of participants completing planned therapy | End of cycle 6 (24 weeks, each cycle is 28 days)
  Number of participants completing the planned six cycles of therapy, along with description of cycle delays
Proportion of participants completing planned therapy | End of cycle 6 (24 weeks, each cycle is 28 days)
  Proportion of participants completing the planned six cycles of therapy, along with description of cycle delays
Disease response rate | End of cycle 6 (24 weeks, each cycle is 28 days)
  Objective disease response rate determined using International Working Group criteria
Decitabine (DAC) incorporation in DNA as AUC | End of cycle 6 (24weeks, each cycle is 28 days)
  Decitabine (DAC) incorporation in DNA of peripheral blood mononuclear cells as measured by mass spectrometry (AZA-MS) and computed as the area under the curve (AUC) per treatment cycle
Global DNA methylation | End of cycle 6 (24weeks, each cycle is 28 days)
  Mean methylcytosine/cytosine ratio in DNA of peripheral blood mononuclear cells within a treatment cycle as measured by mass spectrometry (AZA-MS)
Percentage of Bone Marrow haematopoietic progenitors (HPCs) progressing through the cell cycle | End of cycle 6 (24 weeks, each cycle is 28 days)
  Percentage of Bone Marrow haematopoietic progenitors (HPCs) progressing through the cell cycle as determined by flow cytometry
Percentage of cluster of differentiation 34 (CD34)+ cluster of differentiation 45 (CD45) dimLin- Haematopoietic progenitor cells (HPCs)/ Mononuclear cells (MNCs) per microlitre (uL) of peripheral blood as measured by flow cytometry | End of cycle 6 (24 weeks, each cycle is 28 days)
  Percentage of CD34+CD45dimLin- HPCs /MNCs/uL of peripheral blood as measured by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: John Pimanda, Professor, Principal Investigator — University of New South Wales
Locations (5):
- Australia (5):
  - Prince of Wales Hospital, Sydney, New South Wales
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Concord Repatriation and General Hospital, Sydney, New South Wales
  - Nepean Hospital, Sydney, New South Wales
  - Westmead Hospital, Westmead, New South Wales

IPD SHARING:
Plan to Share IPD: No